CLINICAL TRIAL: NCT03520075
Title: A Phase 1-2 Study of the Safety, Pharmacokinetics, and Activity of ASTX029 in Subjects With Advanced Solid Tumors
Brief Title: Study of ASTX029 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASTX029-01
Record Dates: First submitted 2018-04-18; First posted 2018-05-09 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor, Adult
Keywords: Neoplasms; Solid Tumors; Antineoplastic Agents; MAPK; ERK
MeSH Terms: conditions — Neoplasms | interventions — ASTX029

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Phase 1A: Cohort 1 Dose Escalation (Experimental): Participants received ASTX029 10 milligrams (mg), powder in bottle (PiB), orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fed state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 2 Dose Escalation (Experimental): Participants received ASTX029 20 mg, PiB, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fed state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 3 Dose Escalation (Experimental): Participants received ASTX029 60 mg, PiB, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fed state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 4 Dose Escalation (Experimental): Participants received ASTX029 120 mg, PiB, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fed state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 5 Dose Escalation (Experimental): Participants received ASTX029 200 mg, orally, PiB, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fed state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 6 Dose Escalation (Experimental): Participants received ASTX029 80 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fed state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 7 Dose Escalation (Experimental): Participants received ASTX029 120 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fed state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 8 Dose Escalation (Experimental): Participants received ASTX029 40 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fasted state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 9 Dose Escalation (Experimental): Participants received ASTX029 80 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fasted state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 10 Dose Escalation (Experimental): Participants received ASTX029 120 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fasted state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 11 Dose Escalation (Experimental): Participants received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fasted state.
  Interventions: Drug: ASTX029
- Phase 1A: Cohort 12 Dose Escalation (Experimental): Participants received ASTX029 280 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fasted state.
  Interventions: Drug: ASTX029
- Phase 1B Dose Expansion (Experimental): Participants received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fasted state.
  Interventions: Drug: ASTX029
- Phase 2: Cohort A (Experimental): Participants with neuroblastoma RAS (NRAS)-mutant melanoma received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
  Interventions: Drug: ASTX029
- Phase 2: Cohort B (Experimental): Participants with Kirsten RAS (KRAS)-mutant or KRAS-amplified non-small cell lung cancer (NSCLC) received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
  Interventions: Drug: ASTX029
- Phase 2: Cohort C (Experimental): Participants with B isoform of RAF kinase (BRAF) V600-mutant cancers (non-colorectal cancers) received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
  Interventions: Drug: ASTX029
- Phase 2: Cohort D (Experimental): Participants with BRAF-fusion cancers received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
  Interventions: Drug: ASTX029
- Phase 2: Cohort E (Experimental): Participants with gynecological cancers with alterations in the mitogen-activated protein kinase (MAPK) pathway received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
  Interventions: Drug: ASTX029
- Phase 2: Cohort F (Experimental): Participants with tumors that were characterized by other gene aberrations (that upregulate the MAPK signal pathway) received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
  Interventions: Drug: ASTX029

INTERVENTIONS:
Drug: ASTX029 — PiB
  Arms: Phase 1A: Cohort 1 Dose Escalation; Phase 1A: Cohort 2 Dose Escalation; Phase 1A: Cohort 3 Dose Escalation; Phase 1A: Cohort 4 Dose Escalation; Phase 1A: Cohort 5 Dose Escalation
Drug: ASTX029 — Tablet
  Arms: Phase 1A: Cohort 10 Dose Escalation; Phase 1A: Cohort 11 Dose Escalation; Phase 1A: Cohort 12 Dose Escalation; Phase 1A: Cohort 6 Dose Escalation; Phase 1A: Cohort 7 Dose Escalation; Phase 1A: Cohort 8 Dose Escalation; Phase 1A: Cohort 9 Dose Escalation; Phase 1B Dose Expansion; Phase 2: Cohort A; Phase 2: Cohort B; Phase 2: Cohort C; Phase 2: Cohort D; Phase 2: Cohort E; Phase 2: Cohort F

SUMMARY:
This study is a first-in-human, open-label, multicenter, Phase 1-2 study to assess the safety, pharmacokinetics, pharmacodynamics, and preliminary clinical activity of ASTX029 administered orally to participants with advanced solid malignancies who are not candidates for approved or available therapies.

DETAILED DESCRIPTION:
ASTX029 is a synthetic small molecule inhibitor of extracellular signal-regulated kinases (ERKs) 1/2. ASTX029 has not been previously evaluated in human participants. The Phase 1 portion of this study will assess safety and determine the maximum tolerated dose, the recommended Phase 2 dose (RP2D), and the recommended dosing regimen of ASTX029 administered orally. The Phase 2 portion will assess preliminary clinical activity in tumors characterized by gene aberrations in the mitogen-activated protein kinase (MAPK) signal pathway that may confer sensitivity to ASTX029.

ELIGIBILITY:
Inclusion Criteria:

Participants must fulfill all of the following inclusion criteria.

1. Able to understand and comply with study procedures, understand the risks involved in the study, and provide written informed consent before any study-specific procedure is performed.
2. Men or women 18 years of age or older.
3. Participants with histologically or cytologically confirmed advanced solid tumors that are metastatic or unresectable, who are refractory or have relapsed after treatment with available therapies or for whom standard life-prolonging measures or approved therapies are not available. In Phase 1 Part B and in the Phase 2 portion of the protocol, participants must also have documented gene alterations in the MAPK pathway as detailed in the protocol.
4. In Phase 1 Part B of the protocol, participants must have disease lesions that are amenable to biopsy.
5. In the Phase 2 portion of the protocol, participants must have measurable disease according to RECIST v1.1.
6. Eastern Cooperative Oncology Group performance status 0 to 2.
7. Acceptable organ function as evidenced by the following laboratory data:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase ≤2×upper limit of normal (ULN) or ≤3 ULN in the presence of liver metastases.
   2. Total serum bilirubin ≤1.5×ULN.
   3. Absolute neutrophil count (ANC) ≥1500 cells/mm3.
   4. Platelet count ≥100,000 cells/mm3.
   5. Calculated creatinine clearance (by the standard Cockcroft Gault formula) of ≥50 mL/min or glomerular filtration rate of ≥50 mL/min.
8. Women of child-bearing potential (according to recommendations of the Clinical Trial Facilitation Group [CTFG]; see protocol for details) must not be pregnant or breastfeeding and must have a negative pregnancy test within 24 hours before the first dose of study treatment. While receiving study treatment and for at least 5 half-lives of ASTX029 or metabolite plus 30 days after completing treatment, women of child-bearing potential must agree to practice highly effective contraceptive measures (as described in the protocol) and must refrain from donating eggs (ova, oocytes) for the purpose of reproduction.
9. Men with female partners of child-bearing potential (according to recommendations of the CTFG; see protocol for details) must agree to, during the treatment period and for at least 5 half-lives of ASTX029 or metabolite plus 90 days after completing treatment, practice highly effective contraceptive measures (as described in the protocol), not to father a child, and to refrain from donating sperm.

Exclusion Criteria:

1. Hypersensitivity to ASTX029 or excipients of the drug product.
2. Poor medical risk in the investigator's opinion because of systemic diseases in addition to the cancer under study, for example, uncontrolled infections.
3. Life-threatening illness, significant organ system dysfunction, or other condition that, in the investigator's opinion, could compromise participants safety or the integrity of study outcomes or interfere with the absorption or metabolism of ASTX029.
4. Prior anticancer treatments or therapies within the indicated time window prior to first dose of study treatment (ASTX029), as follows:

   1. Cytotoxic chemotherapy or radiotherapy within 3 weeks prior. Palliative radiotherapy to a single lesion within 2 weeks prior. Any encountered treatment-related toxicities (excepting alopecia) not stabilized or resolved to ≤Grade 1.
   2. Monoclonal antibodies within 4 weeks prior. Any encountered treatment-related toxicities not stabilized or resolved to ≤Grade 1.
   3. Molecularly targeted drug or investigational drugs, without the potential for delayed toxicity, within 4 weeks of the first dose of study treatment or 5 half-lives (minimum 14 days), whichever is shorter. Any encountered treatment-related toxicities (excepting alopecia) not stabilized or resolved to ≤Grade 1.
5. Prior treatment with extracellular signal-regulated kinase (ERK) inhibitors.
6. History of, or at risk for, cardiac disease, as evidenced by 1 or more of the following conditions:

   1. Abnormal left ventricular ejection fraction (LVEF; <50%) on echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan.
   2. Congestive cardiac failure of ≥Grade 3 severity according to New York Heart Association functional classification defined as patients with marked limitation of activity and who are comfortable only at rest.
   3. Unstable cardiac disease including unstable angina or hypertension as defined by the need for overnight hospital admission within the last 3 months (90 days).
   4. History or evidence of long QT interval corrected for heart rate (QTc), ventricular arrhythmias including ventricular bigeminy, complete left bundle branch block, clinically significant bradyarrhythmias such as sick sinus syndrome, second- and third-degree atrioventricular (AV) block, presence of cardiac pacemaker or defibrillator, or other significant arrhythmias.
   5. Screening 12-lead electrocardiogram (ECG) with measurable QTc interval of ≥470 msec. (Fridericia's formula should be used to calculate the QTc interval throughout the study.)
7. Known history of human immunodeficiency virus (HIV) infection or seropositive results consistent with active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection.
8. Known brain metastases, unless previously treated and stable for at least 3 months with or without steroids.
9. Known significant mental illness or other conditions, such as active alcohol or other substance abuse that, in the opinion of the investigator, predispose the participant to high risk of noncompliance with the protocol treatment or assessments.
10. History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including:

    1. Presence of predisposing factors to RVO or CSR (eg, uncontrolled glaucoma or ocular hypertension, uncontrolled diabetes mellitus) or
    2. Visible retinal pathology as assessed by ophthalmic examination at screening that is considered a risk factor for RVO or CSR such as:

       * Evidence of optic disc cupping or
       * Evidence of new visual field defects on automated perimetry or
       * Intraocular pressure >21 mmHg as measured by tonography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (19):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Southern California Norris Comprehensive Cancer Center Site#114, Los Angeles, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute Site# 107, Los Angeles, California
  - Hoag Memorial Hospital Site#115, Newport Beach, California
  - University of California Davis Medical Center Site #121, Sacramento, California
  - California Pacific Medical Center - Sutter Pacific Medical Center Site#117, San Francisco, California
  - Smilow Cancer Hospital at Yale New Haven Site#105, New Haven, Connecticut
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - The Sidney Kimmel Comprehensive Cancer Center Site#106, Baltimore, Maryland
  - Massachusetts General Hospital Site#103, Boston, Massachusetts
  - Dana Farber Cancer Institute Site#104, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center Site #113, Ann Arbor, Michigan
  - Columbia University Irving Medical Center - Herbert Irving Pavilion Site#112, New York, New York
  - Providence Portland Medical Center Site #118, Portland, Oregon
  - Oregon Health and Science University Site #122, Portland, Oregon
  - University of Pennsylvania-Abramson Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center Site#111, Houston, Texas
  - START - South Texas Accelerated Research Therapeutics, LLC Site# 101, San Antonio, Texas
  - Virginia Cancer Specialists Site#102, Fairfax, Virginia
- France (2):
  - Centre Léon Bérard Service d'Oncologie Médicale Site#202, Lyon, Auvergne-Rhône-Alpes
  - Hôpital de la Timone Site #201, Marseille
- Spain (6):
  - Institut Català d'Oncologia Badalona Site#240, Barcelona
  - Hospital Universitari Vall d'Hebrón Servicio de Oncología, Sala coordinación UITM Site#243, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario Dexeus Site#241, Barcelona
  - Clinica Universidad de Navarra Madrid Site #242, Madrid
  - Clínica Universidad de Navarra Site#242, Madrid
- United Kingdom (4):
  - The Christie NHS Foundation Trust Site#220, Manchester, England
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust Site #221, Newcastle upon Tyne
  - Churchill Hospital Site #224, Oxford

REFERENCES:
- [Derived] Munck JM, Berdini V, Bevan L, Brothwood JL, Castro J, Courtin A, East C, Ferraldeschi R, Heightman TD, Hindley CJ, Kucia-Tran J, Lyons JF, Martins V, Muench S, Murray CW, Norton D, O'Reilly M, Reader M, Rees DC, Rich SJ, Richardson CJ, Shah AD, Stanczuk L, Thompson NT, Wilsher NE, Woolford AJ, Wallis NG. ASTX029, a Novel Dual-mechanism ERK Inhibitor, Modulates Both the Phosphorylation and Catalytic Activity of ERK. Mol Cancer Ther. 2021 Oct;20(10):1757-1768. doi: 10.1158/1535-7163.MCT-20-0909. Epub 2021 Jul 30. PMID 34330842

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at regional sites in United States (US), France, Spain, and United Kingdom (UK) from 07 May 2018 to 03 March 2025.
Pre-assignment Details: A total of 192 participants were enrolled in the study to receive ASTX029, of which 2 participants died before receiving treatment. The study was conducted in 2 phases: Phase 1 included Cohorts 1-12 in Part A (Dose Escalation) and a single cohort for Part B (Dose Expansion) and Phase 2 included Cohorts A to F.
Period: Phase 1 (Dose Escalation)
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Started | 3 | 3 | 3 | 5 | 10 | 7 | 3 | 3 | 3 | 3 | 7 | 7 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Safety Analysis Set Included All Participants Who Received Any Amount of Study Drug. | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 7 | 7 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 5 | 10 | 7 | 3 | 3 | 3 | 3 | 6 | 7 | 19 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 3 | 2 | 6 | 5 | 3 | 2 | 3 | 1 | 5 | 7 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Complete Consent Withdrawal | 1 | 0 | 0 | 2 | 3 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 (Dose Expansion)
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 15 | 12 | 9 | 32 | 15
Safety Analysis Set Included All Participants Who Received Any Amount of Study Drug. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 15 | 12 | 9 | 32 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 5 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 15 | 12 | 9 | 27 | 15
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 13 | 9 | 5 | 14 | 12
Not completed — Complete Consent Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 3 | 10 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included data from all participants who received any amount of study drug.
Groups:
- Phase 1A: Cohort 1 Dose Escalation: Participants received ASTX029 10 mg, PiB, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fed state.
- Phase 2: Cohort A: Participants with NRAS-mutant melanoma received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
- Phase 2: Cohort B: Participants with KRAS-mutant or KRAS-amplified NSCLC received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
- Phase 2: Cohort C: Participants with BRAF V600-mutant cancers (non-colorectal cancers) received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
- Phase 2: Cohort E: Participants with gynecological cancers with alterations in the MAPK pathway received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months.
- Total: Total of all reporting groups
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F | Total
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 7 | 7 | 20 | 32 | 15 | 12 | 9 | 32 | 14 | 190
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 | 0 | 2 | 3 | 5 | 5 | 3 | 3 | 1 | 2 | 2 | 4 | 3 | 11 | 14 | 5 | 7 | 3 | 16 | 7 | 96
  65 - 84 | 3 | 1 | 0 | 0 | 5 | 3 | 0 | 2 | 1 | 1 | 3 | 4 | 8 | 18 | 9 | 5 | 6 | 16 | 7 | 92
  >=85 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 5 | 6 | 3 | 3 | 3 | 3 | 1 | 2 | 4 | 12 | 12 | 10 | 7 | 5 | 32 | 6 | 121
  Male | 0 | 1 | 1 | 0 | 4 | 3 | 0 | 0 | 0 | 2 | 5 | 3 | 8 | 20 | 5 | 5 | 4 | 0 | 8 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic, Latino/a, or Spanish origin | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 3 | 3 | 1 | 4 | 2 | 22
  Not of Hispanic, Latino/a, or Spanish origin | 2 | 3 | 3 | 5 | 10 | 5 | 2 | 3 | 1 | 3 | 7 | 6 | 19 | 30 | 12 | 8 | 8 | 25 | 12 | 164
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 6
  American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 8
  Native Hawaiian and Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 1 | 3 | 4 | 9 | 6 | 1 | 3 | 3 | 2 | 6 | 5 | 16 | 20 | 12 | 7 | 6 | 27 | 11 | 145
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 4 | 2 | 4 | 1 | 21
  Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as adverse events (AEs) graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria that occurred during the first cycle of treatment and represented any 1 of the following: grade 4 thrombocytopenia of any duration; ≥grade 3 hematologic toxicity with complications (e.g., grade 3 thrombocytopenia with bleeding or transfusion requirement); febrile neutropenia of any duration or grade 4 neutropenia of 5 days or more duration; liver-associated abnormalities; ≥grade 2 eye disorders; symptomatic grade 2 cutaneous toxicities (including skin rash); any other ≥grade 3 nonhematologic AE except grade 3 nausea, vomiting, or diarrhea; Any event that, in the opinion of the Data and Safety Review Committee (DSRC), would suggest that further dose escalation would put subjects at unacceptable risk.
Time Frame: Cycle 1 (cycle length = 21 days)
Population: The safety analysis set included data from all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 7 | 7 | 20
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Phase 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAEs are defined as events that first occurred or worsened on or after the date of the first dose of study treatment until 30 days after the last dose of study treatment or until the start of a posttreatment alternative anti-cancer treatment, whichever occurs first, with the following exceptions: events that occurred after 30 days beyond the last dose of study treatment or the start of a posttreatment alternative anti-cancer treatment will also be considered treatment-emergent if the events are both serious and related to the study treatment.
Time Frame: From first dose of study drug up to 30 days after last dose (Up to 74 months)
Population: The safety analysis set included data from all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 7 | 7 | 20
Participants | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 7 | 7 | 20

3. Primary Outcome: Phase 2: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: The ORR was calculated as the number of evaluable participants whose best response was complete response (CR) or partial response (PR), divided by the total number of participants evaluable for ORR analysis. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Percentages were rounded off to the nearest single decimal place
Time Frame: Every 2 cycles for the first 4 cycles and then every 4 cycles thereafter until disease progression (Up to 74 months)
Population: The efficacy analysis set included all participants who received any amount of study drug. The ORR analysis was based on participants who were in the efficacy analysis set and who had disease assessment at baseline and at least 1 follow-up disease assessment or participants who died or stopped treatment before the first scheduled disease assessment due to clinical progression or toxicity.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 32 | 15 | 12 | 9 | 32 | 14
percentage of participants | 12.5 [4.4 to 26.4] | 0 [0 to 18.1] | 8.3 [0.4 to 33.9] | 0 [0 to 28.3] | 12.5 [4.4 to 26.4] | 7.1 [0.4 to 29.7]

4. Secondary Outcome: Phase 1: Area Under the Concentration-time Curve From Time Zero to 24 Hours (AUC0-24) of ASTX029
Description: As per planned analysis, data for participants from Part A (Dose Escalation) and Part B (Expansion) were combined for Cohort 11 (200 mg). 2 participants who received 200 and 280 mg respectively, in Cycle 1 Day1 (C1D1), received 120 mg in Cycle 2 and Day 1 (C2D1) and hence counted in Cohort 10. 1 participant who received 280 mg in C1D1, received 200 mg in C2D1 and hence counted in Cohort 11.
Time Frame: Pre-dose on Day 1 of Cycles 1 and 2 and at 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose on Day 1 of Cycles 1 and 2 (Cycle length = 21 days)
Population: The pharmacokinetics (PK) analysis set included all participants who had received study drug with available plasma concentrations and PK parameters for ASTX029. Overall number of participants analyzed is the number of participants with data available for analysis. Number analyzed are unique number of participants out of all the assessed participants with data available at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliters (h*ng/mL)
Groups:
- Phase 1A Cohort 11 Dose Escalation and Phase 1B Dose Expansion: Participants received ASTX029 200 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fasted state.
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A Cohort 11 Dose Escalation and Phase 1B Dose Expansion | Phase 1A: Cohort 12 Dose Escalation
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 2 | 3 | 5 | 26 | 7
hours*nanograms/milliliters (h*ng/mL)
  Cycle 1 Day 1 (C1D1): number analyzed (Participants) | 2 | 3 | 3 | 5 | 10 | 6 | 3 | 2 | 3 | 3 | 26 | 7
  Cycle 1 Day 1 (C1D1) | 277 (20.1) | 361 (222.0) | 1150 (10.0) | 4020 (83.0) | 7250 (63.7) | 1810 (126.9) | 3360 (140.4) | 3080 (128.2) | 6500 (64.3) | 5710 (27.1) | 13400 (46.4) | 17800 (83.6)
  Cycle 2 Day 1 (C2D1): number analyzed (Participants) | 3 | 2 | 3 | 4 | 5 | 4 | 3 | 2 | 3 | 5 | 23 | 3
  Cycle 2 Day 1 (C2D1) | 339 (58.4) | 618 (11.7) | 1410 (61.4) | 3530 (104.5) | 7550 (76.9) | 2490 (108.4) | 3710 (106.0) | 3370 (117.8) | 6430 (71.6) | 7850 (37.1) | 15400 (57.5) | 25600 (91.9)

5. Secondary Outcome: Phase 1: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-last) of ASTX029
Description: As per planned analysis, data for participants from Part A (Dose Escalation) and Part B (Expansion) were combined for Cohort 11 (200 mg). 2 participants who received 200 and 280 mg respectively, in C1D1 received 120 mg in C2D1 and hence counted in Cohort 10. 1 participant who received 280 mg in C1D1, received 200 mg in C2D1 and hence counted in Cohort 11.
Time Frame: as for outcome 4
Population: The PK analysis set included all participants who had received study drug with available plasma concentrations and PK parameters for ASTX029. Overall number of participants analyzed is the number of participants with data available for analysis. Number analyzed are unique number of participants out of all the assessed participants with data available at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A Cohort 11 Dose Escalation and Phase 1B Dose Expansion | Phase 1A: Cohort 12 Dose Escalation
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 5 | 27 | 7
h*ng/mL
  C1D1: number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 27 | 7
  C1D1 | 262 (18.5) | 347 (215.6) | 1140 (10.0) | 4020 (82.9) | 7250 (63.7) | 1740 (137.5) | 3360 (140.4) | 1620 (215.6) | 6450 (65.8) | 5710 (26.9) | 12800 (51.2) | 17800 (83.6)
  C2D1: number analyzed (Participants) | 3 | 3 | 3 | 4 | 5 | 4 | 3 | 2 | 3 | 5 | 25 | 3
  C2D1 | 321 (56.1) | 298 (177.3) | 1410 (61.5) | 3530 (104.5) | 7530 (77.2) | 2430 (116.3) | 3660 (104.2) | 3340 (116.4) | 6450 (72.0) | 7850 (37.1) | 13500 (80.0) | 25300 (93.7)

6. Secondary Outcome: Phase 1: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of ASTX029
Description: As per planned analysis, data for participants from Part A (Dose Escalation) and Part B (Expansion) were combined for Cohort 11 (200 mg). 2 participants who received 200 and 280 mg respectively, in C1D1, received 120 mg in C2D1 and hence counted in Cohort 10. 1 participant who received 280 mg in C1D1, received 200 mg in C2D1 and hence counted in Cohort 11.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A Cohort 11 Dose Escalation and Phase 1B Dose Expansion | Phase 1A: Cohort 12 Dose Escalation
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 9 | 4 | 3 | 2 | 3 | 5 | 25 | 7
h*ng/mL
  C1D1: number analyzed (Participants) | 2 | 3 | 2 | 5 | 9 | 4 | 3 | 2 | 3 | 3 | 25 | 7
  C1D1 | 327 (3.6) | 358 (209.2) | 1150 (14.1) | 4050 (82.5) | 8170 (53.5) | 1180 (112.9) | 3390 (139.3) | 3120 (126.3) | 6520 (66.6) | 5770 (26.7) | 13500 (47.1) | 17900 (83.1)
  C2D1: number analyzed (Participants) | 3 | 2 | 3 | 3 | 5 | 4 | 2 | 2 | 2 | 5 | 25 | 3
  C2D1 | 346 (52.9) | 243 (228.9) | 1430 (60.9) | 5160 (55.0) | 7670 (75.3) | 2470 (116.1) | 3190 (169.8) | 3420 (113.6) | 5590 (101.3) | 7930 (37.2) | 15700 (59.0) | 25600 (92.2)

7. Secondary Outcome: Phase 1: Maximum Observed Plasma Concentration (Cmax) of ASTX029
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- Phase 1A: Cohort 1 Dose Escalation: Participants received ASTX029 10 mg, PiB, orally, once daily, up to median duration of 1.6 months, under fed state.
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A Cohort 11 Dose Escalation and Phase 1B Dose Expansion | Phase 1A: Cohort 12 Dose Escalation
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 5 | 27 | 7
nanograms/milliliter (ng/mL)
  C1D1 | 109 (48.5) | 217 (165.4) | 469 (9.5) | 1650 (56.8) | 1850 (66.7) | 496 (127.7) | 1490 (141.7) | 742 (301.5) | 2840 (30.8) | 2060 (49.5) | 5240 (61.0) | 6040 (58.4)
  C2D1: number analyzed (Participants) | 3 | 3 | 3 | 4 | 5 | 4 | 3 | 2 | 3 | 5 | 25 | 3
  C2D1 | 143 (177.8) | 107 (119.2) | 598 (111.0) | 903 (228.8) | 1830 (177.6) | 641 (91.4) | 1710 (124.4) | 2330 (130.8) | 1860 (55.8) | 2360 (40.9) | 5350 (78.7) | 8070 (50.7)

8. Secondary Outcome: Phase 1: Minimum Plasma Concentration (Cmin) of ASTX029
Description: As per planned analysis, data for participants from Part A (Dose Escalation) and Part B (Expansion) were combined for Cohort 11 (200 mg). 2 participants who received 200 and 280 mg respectively, in C1D1, received 120 mg in C2D1 and hence counted in Cohort 10. 1 participant who received 280 mg in C1D1, received 200 mg in C2D1 and hence counted in Cohort 11. Data for Cmin was calculated and analyzed for C2D1 only.
Time Frame: Pre-dose and at 0.5, 1, 2, 3, 4, 6, and 8 hours post-dose on Day 1 of Cycle 2 (Cycle length = 21 days)
Population: The PK analysis set included all participants who had received study drug with available plasma concentrations and PK parameters for ASTX029. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A Cohort 11 Dose Escalation and Phase 1B Dose Expansion | Phase 1A: Cohort 12 Dose Escalation
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 5 | 4 | 3 | 2 | 3 | 5 | 25 | 3
ng/mL | 4.38 (86.7) | 1.45 (173.2) | 23.4 (127.8) | 19.3 (149.7) | 18.1 (39.7) | 7.88 (79.3) | 68.1 (128.8) | 8.68 (64.0) | 20.1 (114.7) | 85.3 (206.9) | 188 (194.3) | 168 (85.6)

9. Secondary Outcome: Phase 1: Time to Reach Maximum Concentration (Tmax) of ASTX029
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Groups:
- Phase 1a: Cohort 12: Phase 1A: Cohort 12 Dose Escalation Participants received ASTX029 280 mg, tablets, orally, once daily, on Days 1-21 of each 21-day cycle, up to median duration of 1.6 months, under fasted state.
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A Cohort 11 Dose Escalation and Phase 1B Dose Expansion | Phase 1a: Cohort 12
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 5 | 27 | 7
hours
  C1D1: number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 27 | 7
  C1D1 | 1.08 [0.57 to 3.05] | 0.50 [0.50 to 0.58] | 0.55 [0.47 to 0.97] | 0.50 [0.50 to 1.00] | 0.71 [0.43 to 4.08] | 3.03 [1.08 to 5.73] | 1.00 [0.98 to 3.00] | 1.07 [1.00 to 4.02] | 1.00 [0.47 to 1.88] | 1.88 [0.53 to 1.93] | 1.97 [0.50 to 6.00] | 2.03 [1.00 to 4.00]
  C2D1: number analyzed (Participants) | 3 | 3 | 3 | 4 | 5 | 4 | 3 | 2 | 3 | 5 | 25 | 3
  C2D1 | 0.53 [0.50 to 2.20] | 1.00 [0.55 to 1.05] | 0.50 [0.47 to 0.92] | 2.52 [0.92 to 5.7] | 0.55 [0.50 to 1.00] | 2.48 [0.52 to 3.85] | 1.02 [0.50 to 7.53] | 1.52 [1.00 to 2.03] | 3.00 [2.93 to 5.67] | 2.1 [1.08 to 4] | 2.02 [0.92 to 7.52] | 1.90 [0.55 to 3.85]

10. Secondary Outcome: Phase 1: Elimination Half-Life (T1/2) of ASTX029
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A Cohort 11 Dose Escalation and Phase 1B Dose Expansion | Phase 1A: Cohort 12 Dose Escalation
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 9 | 4 | 3 | 2 | 3 | 5 | 25 | 7
hours
  C1D1: number analyzed (Participants) | 2 | 3 | 2 | 5 | 9 | 4 | 3 | 2 | 3 | 3 | 25 | 7
  C1D1 | 2.42 (42.1) | 1.63 (18.7) | 4.42 (1.8) | 3.75 (26.9) | 3.84 (21.8) | 2.08 (102.4) | 4.28 (11.6) | 5.68 (31.7) | 3.30 (74.7) | 4.00 (13.6) | 3.92 (40.9) | 3.71 (32.9)
  C2D1: number analyzed (Participants) | 3 | 2 | 3 | 3 | 5 | 4 | 2 | 2 | 2 | 5 | 21 | 3
  C2D1 | 3.37 (119.7) | 1.85 (64.8) | 4.98 (31.5) | 3.61 (13.5) | 4.11 (15.9) | 2.58 (95.1) | 1.01 (11.6) | 3.13 (276.4) | 4.67 (24.1) | 3.88 (25.6) | 3.80 (47.2) | 1.28 (72.1)

11. Secondary Outcome: Phase 1: Effect of Food on AUC0-24 of ASTX029
Description: The food effect was to be analyzed only for tablet dosage forms. The participants who were administered 80 mg and 120 mg tablets, under both fed and fasted conditions were reported. As 200 mg dose was administered, as tablets, only under fasted conditions, hence food effect was not assessed for 200 mg dose. The statistical comparison between fed and fasted state treatment arm groups of 80 mg and 120 mg doses is reported in this outcome measure for food effect. The 2 participants who received 200 and 280 mg respectively, in C1D1, received 120 mg in C2D1 and hence counted in Cohort 10.
Time Frame: as for outcome 4
Population: The PK analysis set included all participants who had received study drug with available plasma concentrations and PK parameters for ASTX029. The data is reported here for the arm groups of 80 mg and 120 mg, in both fed and fasted to compare food effect. Overall number of participants analyzed is the number of participants with data available for analysis. Number analyzed are unique number of participants out of all the assessed participants with data available at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation
Number analyzed (Participants) | 6 | 3 | 3 | 5
h*ng/mL
  C1D1: number analyzed (Participants) | 6 | 3 | 3 | 3
  C1D1 | 1810 (126.9) | 3360 (140.4) | 6500 (64.3) | 5710 (27.1)
  C2D1: number analyzed (Participants) | 4 | 3 | 3 | 5
  C2D1 | 2490 (108.4) | 3710 (106.0) | 6430 (71.6) | 7850 (37.1)
Statistical Analysis 1: Comparison: Phase 1A: Cohort 6 Dose Escalation vs Phase 1A: Cohort 9 Dose Escalation; Comparison of effect of food on AUC0-24 between Cohort 6 (fed state) and Cohort 9 (fasted state) treatment arm groups of 80 mg ASTX029 in C1D1; Test type: Superiority; Geometric Least Squares Mean (Geo LSM) = 27.8, 90% CI 2-sided [8.50 to 91.2] — Ratio of Geo LSM was calculated for Cohort 6 (fed state) and Cohort 9 (fasted state) treatment arm groups of 80 mg ASTX029
Statistical Analysis 2: Comparison: Phase 1A: Cohort 6 Dose Escalation vs Phase 1A: Cohort 9 Dose Escalation; Comparison of effect of food on AUC0-24 between Cohort 6 (fed state) and Cohort 9 (fasted state) treatment arm groups of 80 mg ASTX029 in C2D1; Test type: Superiority; Geo LSM = 38.8, 90% CI 2-sided [11.4 to 132] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Phase 1A: Cohort 7 Dose Escalation vs Phase 1A: Cohort 10 Dose Escalation; Comparison of effect of food on AUC0-24 between Cohort 7 (fed state) and Cohort 10 (fasted state) treatment arm groups of 120 mg ASTX029 in C1D1; Test type: Superiority; Geo LSM = 58.9, 90% CI 2-sided [15.7 to 222] — Ratio of Geo LSM was calculated for Cohort 7 (fed state) and Cohort 10 (fasted state) treatment arm groups of 120 mg ASTX029
Statistical Analysis 4: Comparison: Phase 1A: Cohort 7 Dose Escalation vs Phase 1A: Cohort 10 Dose Escalation; Comparison of effect of food on AUC0-24 between Cohort 7 (fed state) and Cohort 10 (fasted state) treatment arm groups of 120 mg ASTX029 in C2D1; Test type: Superiority; Geo LSM = 47.2, 90% CI 2-sided [20.7 to 108] — [estimate comment as in outcome 11, analysis 3]

12. Secondary Outcome: Phase 1: Effect of Food on AUC0-inf of ASTX029
Description: as for outcome 11
Time Frame: as for outcome 4
Population: as for outcome 11
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation
Number analyzed (Participants) | 4 | 3 | 3 | 5
h*ng/mL
  C1D1: number analyzed (Participants) | 4 | 3 | 3 | 3
  C1D1 | 1180 (112.9) | 3390 (139.3) | 6520 (66.6) | 5770 (26.7)
  C2D1: number analyzed (Participants) | 4 | 2 | 2 | 5
  C2D1 | 2470 (116.1) | 3190 (169.8) | 5590 (101.3) | 7930 (37.2)
Statistical Analysis 1: Comparison: Phase 1A: Cohort 6 Dose Escalation vs Phase 1A: Cohort 9 Dose Escalation; Comparison of effect of food on AUC0-inf between Cohort 6 (fed state) and Cohort 9 (fasted state) treatment arm groups of 80 mg ASTX029 in C1D1; Test type: Superiority; Geo LSM = 18.1, 90% CI 2-sided [5.28 to 61.9] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Phase 1A: Cohort 6 Dose Escalation vs Phase 1A: Cohort 9 Dose Escalation; Comparison of effect of food on AUC0-inf between Cohort 6 (fed state) and Cohort 9 (fasted state) treatment arm groups of 80 mg ASTX029 in C2D1; Test type: Superiority; Geo LSM = 44.1, 90% CI 2-sided [8.32 to 234] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Phase 1A: Cohort 7 Dose Escalation vs Phase 1A: Cohort 10 Dose Escalation; Comparison of effect of food on AUC0-inf between Cohort 7 (fed state) and Cohort 10 (fasted state) treatment arm groups of 120 mg ASTX029 in C1D1; Test type: Superiority; Geo LSM = 58.7, 90% CI 2-sided [15.7 to 220] — [estimate comment as in outcome 11, analysis 3]
Statistical Analysis 4: Comparison: Phase 1A: Cohort 7 Dose Escalation vs Phase 1A: Cohort 10 Dose Escalation; Comparison of effect of food on AUC0-inf between Cohort 7 (fed state) and Cohort 10 (fasted state) treatment arm groups of 120 mg ASTX029 in C2D1; Test type: Superiority; Geo LSM = 40.2, 90% CI 2-sided [14.3 to 113] — [estimate comment as in outcome 11, analysis 3]

13. Secondary Outcome: Phase 1: Effect of Food on Cmax of ASTX029
Description: as for outcome 11
Time Frame: as for outcome 4
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation
Number analyzed (Participants) | 6 | 3 | 3 | 5
ng/mL
  C1D1: number analyzed (Participants) | 6 | 3 | 3 | 3
  C1D1 | 496 (127.7) | 1490 (141.7) | 2840 (30.8) | 2060 (49.5)
  C2D1: number analyzed (Participants) | 4 | 3 | 3 | 5
  C2D1 | 641 (91.4) | 1710 (124.4) | 1860 (55.8) | 2360 (40.9)
Statistical Analysis 1: Comparison: Phase 1A: Cohort 6 Dose Escalation vs Phase 1A: Cohort 9 Dose Escalation; Comparison of effect of food on Cmax between Cohort 6 (fed state) and Cohort 9 (fasted state) treatment arm groups of 80 mg ASTX029 in C1D1; Test type: Superiority; Geo LSM = 17.5, 90% CI 2-sided [5.62 to 54.3] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Phase 1A: Cohort 6 Dose Escalation vs Phase 1A: Cohort 9 Dose Escalation; Comparison of effect of food on Cmax between Cohort 6 (fed state) and Cohort 9 (fasted state) treatment arm groups of 80 mg ASTX029 in C2D1; Test type: Superiority; Geo LSM = 34.5, 90% CI 2-sided [12.0 to 99.4] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Phase 1A: Cohort 7 Dose Escalation vs Phase 1A: Cohort 10 Dose Escalation; Comparison of effect of food on Cmax between Cohort 7 (fed state) and Cohort 10 (fasted state) treatment arm groups of 120 mg ASTX029 in C1D1; Test type: Superiority; Geo LSM = 72.6, 90% CI 2-sided [17.6 to 299] — [estimate comment as in outcome 11, analysis 3]
Statistical Analysis 4: Comparison: Phase 1A: Cohort 7 Dose Escalation vs Phase 1A: Cohort 10 Dose Escalation; [analysis description as in outcome 13, analysis 3]; Test type: Superiority; Geo LSM = 72.5, 90% CI 2-sided [29.1 to 181] — [estimate comment as in outcome 11, analysis 3]

14. Secondary Outcome: Phase 1: Effect of Food on Tmax of ASTX029
Description: as for outcome 11
Time Frame: as for outcome 4
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation
Number analyzed (Participants) | 6 | 3 | 3 | 5
hours
  C1D1: number analyzed (Participants) | 6 | 3 | 3 | 3
  C1D1 | 3.03 [1.08 to 5.73] | 1.00 [0.98 to 3.00] | 1.00 [0.47 to 1.88] | 1.88 [0.53 to 1.93]
  C2D1: number analyzed (Participants) | 4 | 3 | 3 | 5
  C2D1 | 2.48 [0.52 to 3.85] | 1.02 [0.50 to 7.53] | 3.00 [2.93 to 5.67] | 2.1 [1.08 to 4]
Statistical Analysis 1: Comparison: Phase 1A: Cohort 6 Dose Escalation vs Phase 1A: Cohort 9 Dose Escalation; Comparison of effect of food on Tmax between Cohort 6 (fed state) and Cohort 9 (fasted state) treatment arm groups of 80 mg ASTX029 in C1D1; Test type: Superiority; p = 0.0388671, Wilcoxon (Mann-Whitney); Hodges-Lehmann Estimator = -2.275, 90% CI 2-sided [-5.2160 to -0.0830] — The Hodges-Lehmann estimator and 90% confidence interval (CI) was calculated using the Moses approximation
Statistical Analysis 2: Comparison: Phase 1A: Cohort 6 Dose Escalation vs Phase 1A: Cohort 9 Dose Escalation; Comparison of effect of food on Tmax between Cohort 6 (fed state) and Cohort 9 (fasted state) treatment arm groups of 80 mg ASTX029 in C2D1; Test type: Superiority; p = 0.4795001, Wilcoxon (Mann-Whitney); Hodges-Lehmann Estimator = 1.45, 90% CI 2-sided [-0.9170 to 5.1500] — The Hodges-Lehmann estimator and 90% CI was calculated using the Moses approximation
Statistical Analysis 3: Comparison: Phase 1A: Cohort 7 Dose Escalation vs Phase 1A: Cohort 10 Dose Escalation; Comparison of effect of food on Tmax between Cohort 7 (fed state) and Cohort 10 (fasted state) treatment arm groups of 120 mg ASTX029 in C1D1; Test type: Superiority; p = 0.8272593, Wilcoxon (Mann-Whitney); Hodges-Lehmann Estimator = -0.45, 90% CI 2-sided [-2.4670 to 0.9500] — The Hodges-Lehmann estimator and 90% CI was calculated using the Moses approximation
Statistical Analysis 4: Comparison: Phase 1A: Cohort 7 Dose Escalation vs Phase 1A: Cohort 10 Dose Escalation; Comparison of effect of food on Tmax between Cohort 7 (fed state) and Cohort 10 (fasted state) treatment arm groups of 120 mg ASTX029 in C2D1; Test type: Superiority; p = 0.5126908, Wilcoxon (Mann-Whitney); Hodges-Lehmann Estimator = 0.583, 90% CI 2-sided [-6.4500 to 3.5000] — The Hodges-Lehmann estimator and 90% CI was calculated using the Moses approximation

15. Secondary Outcome: Phase 1: Inhibition of Phosphorylated Ribosomal S6 Kinase (pRSK) Protein in Response to ASTX029 Treatment in Tumor Biopsies as Assessed by H Score
Description: The protein expression level is quantified through the H-score, calculated from staining intensity within the target cell region. H-Score = (3x % of cells with staining graded 3) + (2x % of cells with staining graded 2) + % of cells with staining graded 1. H-Score ranges between 0 to 300. The H-score is for sum of cytoplasmic H-Score (C pRSK H-Score) and nuclear H-Scores (N pRSK H-Score). C pRSK H-Scores, and nuclear H-Scores were combined to give a single H-score.
Time Frame: 4 hours post-dose on Day 8 of Cycle 2 (Cycle length = 21 days)
Population: Pharmacodynamics analysis set included in the pharmacodynamic and biomarker analyses if they have received study drug and their samples were successfully collected and analyzed. Overall number of participants analyzed is the number of participants with data available for analysis. The data for this outcome measure was collected and analyzed for Phase 1B Dose Expansion cohort only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1B Dose Expansion
Number analyzed (Participants) | 8
score on a scale | 181.6 (172.31)

16. Secondary Outcome: Phase 1: Progression Free Survival (PFS)
Description: The PFS was defined as the number of months from the start of the study treatment to disease progression or death, whichever occurs first. The PFS was analyzed using a Kaplan-Meier method, with PFS time being censored on the date of the last disease assessment. The 90% CI for median PFS was provided using the Kaplan-Meier procedure.
Time Frame: Every 2 cycles for the first 4 cycles and then every 4 cycles thereafter until disease progression (Up to 82 months)
Population: The efficacy analysis set included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 7 | 7 | 20
months | 1.3 [1.2 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 1.2 [1.2 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 8.1 [2.7 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 2.0 [1.1 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 1.2 [0.2 to 4.8] | 1.3 [0.9 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 3.0 [1.2 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 1.1 [1.0 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 1.3 [1.0 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 2.3 [1.4 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 3.0 [0.7 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 2.5 [0.4 to 4.0] | 1.4 [1.2 to 4.2]

17. Secondary Outcome: Phase 1: Overall Survival (OS)
Description: The OS was defined as the number of months from the day the participant was randomized to the date of death (regardless of cause). Participants without a documented death date were censored on the last date they were known to be alive. The OS was presented using a Kaplan-Meier estimate.
  The 90% CI for median OS was provided using the Kaplan-Meier procedure.
Time Frame: Up to 82 months
Population: The efficacy analysis set included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 7 | 7 | 20
months | 13.5 [4.4 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 4.5 [3.4 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 10.2 [4.1 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 3.8 [2.1 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 2.1 [0.5 to 25.5] | 11.3 [4.8 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 8.7 [2.6 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 2.0 [1.1 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 10.9 [1.3 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | NA [NA to NA] — Median was not reached. The lower limit and upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 14.8 [2.7 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 2.5 [1.2 to 13.1] | 15.1 [2.7 to 26.3]

18. Secondary Outcome: Phase 1: Disease Control Rate (DCR)
Description: DCR was calculated as the number of participants whose best response was CR, PR, or stable disease (SD), divided by the total number of participants evaluable for DCR analysis. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. PR was defined as at least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable disease was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. Percentages were rounded off to the nearest single decimal place.
Time Frame: Every 2 cycles for the first 4 cycles and then every 4 cycles thereafter until disease progression (Up to 82 months)
Population: The efficacy analysis set included all participants who received any amount of study drug. The DCR analysis was based on participants who were in the efficacy analysis set and who had disease assessment at baseline and at least 1 follow-up disease assessment or participants who died or stopped treatment before the first scheduled disease assessment due to clinical progression or toxicity.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 10 | 6 | 3 | 3 | 3 | 3 | 7 | 7 | 20
percentage of participants | 0 [0 to 63.2] | 0 [0 to 63.2] | 100 [36.8 to 100] | 40.0 [7.6 to 81.1] | 20.0 [3.7 to 50.7] | 16.7 [0.9 to 58.2] | 66.7 [13.5 to 98.3] | 33.3 [1.7 to 86.5] | 33.3 [1.7 to 86.5] | 33.3 [1.7 to 86.5] | 85.7 [47.9 to 99.3] | 42.9 [12.9 to 77.5] | 30.0 [14 to 50.8]

19. Secondary Outcome: Phase 1: Duration of Response (DoR)
Description: Duration of response was calculated for all responders from the date of the earliest assessment of CR or PR to the date of relapse or death, whichever occurred earlier, or the last disease assessment date for participants without a relapse or death. Duration of SD was calculated for participants whose best response is CR, PR, or SD from the day study drug was first taken to the date of disease progression or death, whichever occurred earlier, or the last disease assessment for participants without disease progression or death.
Time Frame: Every 2 cycles for the first 4 cycles and then every 4 cycles thereafter until disease progression (Up to 82 months)
Population: The efficacy analysis set included all participants who received any amount of study drug. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
days |  |  |  |  |  |  |  |  |  | 484.0 [484.0 to 484.0] | 61.0 [61.0 to 61.00] |  | 252.50 [252.0 to 253.0]

20. Secondary Outcome: Phase 2: AUC0-24 of ASTX029
Time Frame: Pre-dose on Day 1 of Cycles 1, and 3; at 0.5,1, 2, 3, 4, 6, and 8 hours post-dose on Day 1 of Cycle 1, and at 0.5,1, 2, 4, and 8 hours post-dose on Day 1 of Cycle 3 (Cycle length = 21 days)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 24 | 13 | 9 | 9 | 28 | 12
h*ng/mL
  C1D1 | 12200 (69.1) | 13000 (57.2) | 9570 (80.3) | 8730 (100.0) | 12000 (83.3) | 13400 (71.3)
  Cycle 3 Day 1 (C3D1): number analyzed (Participants) | 15 | 4 | 1 | 4 | 16 | 5
  Cycle 3 Day 1 (C3D1) | 11600 (76.1) | 27600 (47.3) | 11500 (NA) — Geometric coefficient of variation was not estimable due to low number of participants at specified time point. | 12800 (36.2) | 12300 (88.7) | 15300 (52.4)

21. Secondary Outcome: Phase 2: AUC0-last of ASTX029
Time Frame: as for outcome 20
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 32 | 15 | 12 | 9 | 32 | 14
h*ng/mL
  C1D1 | 12300 (70.4) | 15000 (68.5) | 7800 (81.7) | 8730 (100.0) | 11500 (80.3) | 12700 (66.9)
  C3D1: number analyzed (Participants) | 19 | 7 | 5 | 5 | 20 | 5
  C3D1 | 8090 (214.2) | 13600 (114.5) | 1960 (369.9) | 11700 (31.5) | 10400 (86.4) | 14000 (52.1)

22. Secondary Outcome: Phase 2: AUC0-inf of ASTX029
Description: Data for Auc0-inf was collected and analyzed for C1D1 only.
Time Frame: Pre-dose on Day 1 of Cycle 1; and at 0.5,1, 2, 3, 4, 6, and 8 hours post-dose on Day 1 of Cycle 1 (Cycle length = 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 28 | 13 | 6 | 7 | 30 | 13
h*ng/mL | 12500 (66.6) | 17100 (60.4) | 10700 (103.0) | 11800 (62.5) | 12500 (74.5) | 13300 (67.5)

23. Secondary Outcome: Phase 2: Cmax of ASTX029
Time Frame: as for outcome 20
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 32 | 15 | 12 | 9 | 32 | 14
ng/mL
  C1D1 | 4430 (70.9) | 5930 (81.3) | 2890 (97.7) | 2840 (239.4) | 4660 (113.6) | 5620 (65.7)
  C3D1: number analyzed (Participants) | 19 | 7 | 5 | 5 | 20 | 5
  C3D1 | 3280 (179.3) | 4730 (150.7) | 780 (464.1) | 5090 (43.5) | 4410 (110.4) | 4860 (66.8)

24. Secondary Outcome: Phase 2: Cmin of ASTX029
Description: Data for Cmin was calculated and analyzed for C3D1 only.
Time Frame: Pre-dose on Day 1 of Cycle 3; and at 0.5,1, 2, 4, and 8 post-dose on Day 1 of Cycle 3 (Cycle length = 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 19 | 7 | 5 | 5 | 20 | 5
ng/mL | 189 (181.0) | 260 (95.5) | 81.7 (102.0) | 144 (78.2) | 205 (104.9) | 246 (67.6)

25. Secondary Outcome: Phase 2: Tmax of ASTX029
Time Frame: as for outcome 20
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 32 | 15 | 12 | 9 | 32 | 14
hours
  C1D1 | 2.03 [0.50 to 4.08] | 1.95 [0.95 to 6.08] | 2.90 [0.50 to 7.55] | 2.07 [0.92 to 7.90] | 2.00 [0.40 to 4.07] | 2.00 [1.00 to 3.87]
  C3D1: number analyzed (Participants) | 19 | 7 | 5 | 5 | 20 | 5
  C3D1 | 2.00 [0.97 to 4.05] | 2.03 [0.58 to 4.05] | 2.03 [0.67 to 7.53] | 1.90 [1.00 to 2.00] | 2.00 [0.48 to 4.17] | 1.97 [0.95 to 4.00]

26. Secondary Outcome: Phase 2: T1/2 of ASTX029
Description: Data for T1/2 was collected and analyzed for C1D1 only.
Time Frame: Pre-dose on Day 1 of Cycle 1; at 0.5,1, 2, 3, 4, 6, and 8 hours post-dose on Day 1 of Cycle 1 (Cycle length = 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 28 | 13 | 6 | 7 | 30 | 13
hours | 2.68 (68.8) | 3.45 (52.0) | 3.79 (19.1) | 3.73 (12.2) | 3.64 (43.2) | 3.39 (48.2)

27. Secondary Outcome: Phase 2: Progression Free Survival
Description: as for outcome 16
Time Frame: Every 2 cycles for the first 4 cycles and then every 4 cycles thereafter until disease progression (Up to 82 months)
Population: The efficacy analysis set included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 32 | 15 | 12 | 9 | 32 | 14
months | 2.8 [1.5 to 5.5] | 2.8 [0.9 to 4.6] | 1.7 [0.8 to 6.1] | 8.0 [1.0 to 9.6] | 3.5 [2.2 to 6.2] | 2.0 [1.2 to 5.5]

28. Secondary Outcome: Phase 2: Overall Survival
Description: The OS was defined as the number of months from the day the participant was randomized to the date of death (regardless of cause). Participants without a documented death date were censored on the last date they were known to be alive. The OS was presented using a KM estimate. The 90% CI for median OS was provided using the Kaplan-Meier procedure.
Time Frame: Up to 82 months
Population: The efficacy analysis set included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 32 | 15 | 12 | 9 | 32 | 14
months | 8.0 [4.4 to 13.6] | 4.9 [1.5 to 10.1] | 6.1 [1.1 to 19.3] | 11.6 [2.0 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 11.2 [6.8 to NA] — Upper limit of 95% CI was not estimable because there was no event time for which the upper bound of the CI for the Kaplan-Meier estimate was less than 0.5. | 9.9 [3.5 to 15.9]

29. Secondary Outcome: Phase 2: Disease Control Rate
Description: DCR was calculated as the number of participants whose best response was CR, PR, or SD, divided by the total number of participants evaluable for DCR analysis. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to <10 mm. PR was defined as at least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable disease was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Every 2 cycles for the first 4 cycles and then every 4 cycles thereafter until disease progression (Up to 82 months)
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 32 | 15 | 12 | 9 | 32 | 14
percentage of participants | 65.6 [49.6 to 79.4] | 60.0 [36 to 80.9] | 41.7 [18.1 to 68.5] | 77.8 [45 to 95.9] | 68.8 [52.8 to 82] | 42.9 [20.6 to 67.5]

30. Secondary Outcome: Phase 2: Duration of Response
Description: as for outcome 19
Time Frame: Every 2 cycles for the first 4 cycles and then every 4 cycles thereafter until disease progression (Up to 82 months)
Population: as for outcome 19
Measure: Median (Full Range); unit: days
Arm/Group | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
Number analyzed (Participants) | 4 | 0 | 1 | 0 | 4 | 1
days | 193.00 [65.0 to 219.0] |  | 144.00 [144.00 to 144.00] |  | 189.50 [102.0 to 260.0] | 750.00 [750.00 to 750.00]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of the study (Up to 82 months)
Description: The Safety Analysis Set included data from all participants who received any amount of study drug.
Arm/Group | Phase 1A: Cohort 1 Dose Escalation | Phase 1A: Cohort 2 Dose Escalation | Phase 1A: Cohort 3 Dose Escalation | Phase 1A: Cohort 4 Dose Escalation | Phase 1A: Cohort 5 Dose Escalation | Phase 1A: Cohort 6 Dose Escalation | Phase 1A: Cohort 7 Dose Escalation | Phase 1A: Cohort 8 Dose Escalation | Phase 1A: Cohort 9 Dose Escalation | Phase 1A: Cohort 10 Dose Escalation | Phase 1A: Cohort 11 Dose Escalation | Phase 1A: Cohort 12 Dose Escalation | Phase 1B Dose Expansion | Phase 2: Cohort A | Phase 2: Cohort B | Phase 2: Cohort C | Phase 2: Cohort D | Phase 2: Cohort E | Phase 2: Cohort F
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 3/3 | 3/5 | 9/10 | 4/6 | 3/3 | 3/3 | 3/3 | 1/3 | 5/7 | 7/7 | 13/20 | 23/32 | 13/15 | 10/12 | 5/9 | 14/32 | 11/14
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 2/3 | 2/5 | 7/10 | 1/6 | 2/3 | 0/3 | 1/3 | 1/3 | 3/7 | 1/7 | 9/20 | 11/32 | 5/15 | 4/12 | 3/9 | 12/32 | 4/14
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 5/5 | 8/10 | 6/6 | 3/3 | 3/3 | 3/3 | 3/3 | 7/7 | 7/7 | 20/20 | 31/32 | 15/15 | 12/12 | 9/9 | 32/32 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1A: Cohort 1 Dose Escalation (N=3) | Phase 1A: Cohort 2 Dose Escalation (N=3) | Phase 1A: Cohort 3 Dose Escalation (N=3) | Phase 1A: Cohort 4 Dose Escalation (N=5) | Phase 1A: Cohort 5 Dose Escalation (N=10) | Phase 1A: Cohort 6 Dose Escalation (N=6) | Phase 1A: Cohort 7 Dose Escalation (N=3) | Phase 1A: Cohort 8 Dose Escalation (N=3) | Phase 1A: Cohort 9 Dose Escalation (N=3) | Phase 1A: Cohort 10 Dose Escalation (N=3) | Phase 1A: Cohort 11 Dose Escalation (N=7) | Phase 1A: Cohort 12 Dose Escalation (N=7) | Phase 1B Dose Expansion (N=20) | Phase 2: Cohort A (N=32) | Phase 2: Cohort B (N=15) | Phase 2: Cohort C (N=12) | Phase 2: Cohort D (N=9) | Phase 2: Cohort E (N=32) | Phase 2: Cohort F (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intracranial mass (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal stoma output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1A: Cohort 1 Dose Escalation (N=3) | Phase 1A: Cohort 2 Dose Escalation (N=3) | Phase 1A: Cohort 3 Dose Escalation (N=3) | Phase 1A: Cohort 4 Dose Escalation (N=5) | Phase 1A: Cohort 5 Dose Escalation (N=10) | Phase 1A: Cohort 6 Dose Escalation (N=6) | Phase 1A: Cohort 7 Dose Escalation (N=3) | Phase 1A: Cohort 8 Dose Escalation (N=3) | Phase 1A: Cohort 9 Dose Escalation (N=3) | Phase 1A: Cohort 10 Dose Escalation (N=3) | Phase 1A: Cohort 11 Dose Escalation (N=7) | Phase 1A: Cohort 12 Dose Escalation (N=7) | Phase 1B Dose Expansion (N=20) | Phase 2: Cohort A (N=32) | Phase 2: Cohort B (N=15) | Phase 2: Cohort C (N=12) | Phase 2: Cohort D (N=9) | Phase 2: Cohort E (N=32) | Phase 2: Cohort F (N=14)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 2 | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 3 | 7 | 9 | 3 | 5 | 2 | 14 | 5
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyschromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 5 | 0 | 0 | 1 | 4 | 4
Visual field defect (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Macular detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 0 | 1 | 3 | 2
Central serous chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Presbyopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual brightness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 4 | 1 | 2 | 2 | 1 | 2 | 3 | 3 | 7 | 10 | 8 | 5 | 4 | 15 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 3 | 4 | 10 | 19 | 6 | 5 | 6 | 23 | 8
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 5 | 2 | 0 | 2 | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 5 | 9 | 0 | 0 | 3 | 1 | 2
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 3 | 1 | 6 | 6 | 4 | 5 | 2 | 13 | 3
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 1 | 0 | 1 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 5 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 2 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 3 | 1
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 1 | 0 | 1 | 2 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 2 | 1
Fatigue (General disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 5 | 3 | 7 | 10 | 4 | 3 | 5 | 15 | 6
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 5 | 2 | 0 | 0 | 2 | 1
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 5 | 1 | 1 | 2 | 6 | 3
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 4 | 1 | 0 | 0 | 7 | 2
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Injection site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 2 | 1
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 5 | 2 | 0 | 1 | 0 | 2 | 2 | 1 | 2 | 6 | 0 | 0 | 0 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 5 | 1 | 0 | 0 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 0 | 2 | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 2 | 2 | 1
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 2 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood corticotrophin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 6 | 5 | 2 | 2 | 9 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 6 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 0 | 1 | 1 | 5 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 3 | 1 | 2 | 1 | 0 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 3 | 1 | 1 | 5 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 7 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 1 | 1 | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 1 | 1 | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 0 | 0 | 0 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 1 | 4 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 2 | 2 | 3 | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 2 | 3 | 1 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 4 | 4 | 4 | 0 | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 4 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 7 | 1 | 0 | 0 | 4 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 6 | 4 | 2 | 1 | 9 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 4 | 6 | 2 | 0 | 0 | 3 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Skin indentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Venous injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The ASTX029 clinical development program was terminated by the sponsor due to the changing treatment landscape.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03520075/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT03520075/SAP_001.pdf